CLINICAL TRIAL: NCT05850377
Title: 5-Aminolevulinic Acid (5-ALA) Gliolan®: Usage Increase Proposal for Neurosurgical Procedures in High-Grade Gliomas
Status: Not yet recruiting | Type: Observational
Sponsor: Sociedad de Lucha Contra el Cáncer del Ecuador (Other)
Responsible Party: Sponsor
Other Study IDs: CISOLGYE20230023
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: High Grade Glioma; Glioma; Glioma, Malignant; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Photosensitizing Agents; Neoplasm Malignant; Brain Neoplasms, Adult, Malignant; Central Nervous System Neoplasms; Brain Tumor; Tumour, Residual
Keywords: High Grade Glioma; 5-ALA; Aminolevulinic Acid; Malignant Glioma; Photodynamic Therapy; Fluorescence-guided Surgery; Photosensitizing Agents; Tumor Resection
MeSH Terms: conditions — Glioma; Neoplasms, Neuroepithelial; Neuroectodermal Tumors; Neoplasms; Brain Neoplasms; Central Nervous System Neoplasms; Neoplasm, Residual | interventions — Aminolevulinic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with known or suspected High-Grade Gliomas: Patients with malignant gliomas undergoing neurosurgical procedures using 5-aminolevulinic acid (5-ALA)-based photodynamic therapy
  Interventions: Drug: 5-Aminolevulinic Acid (5-ALA) Gliolan®; Procedure: Fluorescence-Guided Surgery using 5-aminolevulinic acid (5-ALA)

INTERVENTIONS:
Drug: 5-Aminolevulinic Acid (5-ALA) Gliolan® — Gliolan® is presented as a powder for oral solution in 60 ml colorless glass vials and is administered orally three hours (range 2-4 hours) before anaesthesia. One bottle contains 1.17 g of 5-aminolevulinic acid (5-ALA), corresponding to 1.5 g 5-aminolevulinic acid hydrochloride (5-ALA HCl). The recommended dose is 20 mg 5-ALA HCl per kilogram body weight. One ml of reconstituted solution contains 23.4 mg of 5-ALA, corresponding to 30 mg 5-ALA HCl.
  Other Names: Gliolan®; Gleolan®
Procedure: Fluorescence-Guided Surgery using 5-aminolevulinic acid (5-ALA) — During the surgical exploration of the glioma, the neurosurgeon will attempt to identify the mass. The location of the tumor will be assessed using the blue-light filtered microscope. A biopsy of the fluorescent region will be taken to confirm the glioma subtype. The tumor will then be maximally resected.

SUMMARY:
The goal of this observational study is to evaluate disease-free survival (DFS) in patients with malignant gliomas undergoing neurosurgical procedures using 5-aminolevulinic acid (5-ALA)-based photodynamic therapy

DETAILED DESCRIPTION:
The investigators are proposing a study that provides descriptive understanding of patients with High-Grade Gliomas in Ecuador. The primary objective of this pilot study is to lay the foundations for the development of a multicenter registry patients with malignant gliomas undergoing neurosurgical procedures using 5-aminolevulinic acid (5-ALA)-based photodynamic therapy, which will provide high-quality real data and serve as a basis for the application to future projects and elaboration of public policies in the medium and long term.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years (in pediatric cases will be included in the Central Nervous System (CNS) tumor board to make decisions on therapeutic management)
* Patients with radiological suspicion (contrast uptake) of high-grade glioma (Grade III-IV)
* Patients with high-grade and residual glioma following surgery for gross total resection
* Patients with recurrent gliomas with reoperation criteria who previously received radiotherapy and chemotherapy
* Patients for whom at least one postoperative magnetic resonance imaging (MRI) was available (up to 28 days after surgery and strictly before the start of radiotherapy)
* Progressing, low-grade infiltrative gliomas with one of the following criteria:
* Anaplastic foci with contrast uptake in MRI
* Spectroscopy study in anaplastic suspected area with high malignancy criteria
* Positive choline PET-CT (positron emission tomography / computer tomography)

Exclusion Criteria:

* Tumors extending across midline
* Basal ganglia tumor
* Brainstem tumor
* Multifocal gliomas
* Suspected low-grade glioma without anaplastic foci
* Neuraxial dissemination (ependymoma)
* Karnofsky grade less than 60%
* Infants or pregnant women
* Acute or chronic types of porphyria
* Non-acceptance of Fluorescence-Guided Surgery
* Renal insufficiency confirmed by nephrological assessment
* Hepatic impairment confirmed by gastroenterological assessment
* Severe heart disease confirmed by cardiological assessment
* Decompensated diabetes confirmed by endocrinological assessment
* Known allergy to any contrast agent and/or previous history of anaphylactic shock
* Hypersensitivity to the active substance or porphyrins
* Asthma confirmed by pulmonological assessment
* Pacemaker use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-Grade Gliomas patients according to the 2021 World Health Organization (WHO) classification at Instituto Oncológico Nacional Dr. Juan Tanca Marengo
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free-Survival (PFS) | 36 months
  Disease-Free-Survival calculates the time from treatment until the recurrence of disease or death after undergoing Fluorescence-Guided Surgery using 5-aminolevulinic acid (5-ALA)

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  Overall survival is defined as time from initiation to death of any cause
Quality of life as measured by the Functional Assessment of Cancer Therapy - Brain (FACT-Br) questionnaire | 36 months
  The questionnaire provides an additional set of disease-specific questions pertaining to brain neoplasms. It consists of 46 items that refer to general issues of quality of life and specific to tumor location. Possible scores range from 0 to 108, with higher scores indicating better quality of life.
Average length of hospital stay (ALOS) | 36 months
  The average length of stay in hospitals is often used as an indicator of efficiency. The ALOS refers to the average number of days that patients spend in hospital after surgery. It is calculated by dividing the number of bed-days by the number of discharges after procedure. Average length of stay range from 1 day to 4.5 days. Longer than average stays are usually a symptom of poor communication, quality of care, and effectiveness of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Valarezo Chuchuca, MD, Principal Investigator — Sociedad de Lucha Contra el Cáncer del Ecuador
Locations (1):
- Sociedad de Lucha Contra el Cáncer, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Widhalm G, Minchev G, Woehrer A, Preusser M, Kiesel B, Furtner J, Mert A, Di Ieva A, Tomanek B, Prayer D, Marosi C, Hainfellner JA, Knosp E, Wolfsberger S. Strong 5-aminolevulinic acid-induced fluorescence is a novel intraoperative marker for representative tissue samples in stereotactic brain tumor biopsies. Neurosurg Rev. 2012 Jul;35(3):381-91; discussion 391. doi: 10.1007/s10143-012-0374-5. Epub 2012 Mar 10. PMID 22407140
- [Background] Nitta T, Sato K. Prognostic implications of the extent of surgical resection in patients with intracranial malignant gliomas. Cancer. 1995 Jun 1;75(11):2727-31. doi: 10.1002/1097-0142(19950601)75:113.0.co;2-h. PMID 7743477
- [Background] Lacroix M, Abi-Said D, Fourney DR, Gokaslan ZL, Shi W, DeMonte F, Lang FF, McCutcheon IE, Hassenbusch SJ, Holland E, Hess K, Michael C, Miller D, Sawaya R. A multivariate analysis of 416 patients with glioblastoma multiforme: prognosis, extent of resection, and survival. J Neurosurg. 2001 Aug;95(2):190-8. doi: 10.3171/jns.2001.95.2.0190. PMID 11780887
- [Background] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043
- [Background] Inoue T, Endo T, Nagamatsu K, Watanabe M, Tominaga T. 5-aminolevulinic acid fluorescence-guided resection of intramedullary ependymoma: report of 9 cases. Neurosurgery. 2013 Jun;72(2 Suppl Operative):ons159-68; discussion ons168. doi: 10.1227/NEU.0b013e31827bc7a3. PMID 23149963
- [Background] Eicker SO, Floeth FW, Kamp M, Steiger HJ, Hanggi D. The impact of fluorescence guidance on spinal intradural tumour surgery. Eur Spine J. 2013 Jun;22(6):1394-401. doi: 10.1007/s00586-013-2657-0. Epub 2013 Jan 10. PMID 23307195
- [Background] Beez T, Sarikaya-Seiwert S, Steiger HJ, Hanggi D. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of brain tumors in children--a technical report. Acta Neurochir (Wien). 2014 Mar;156(3):597-604. doi: 10.1007/s00701-014-1997-9. Epub 2014 Jan 22. PMID 24449149
- [Background] Eicker S, Sarikaya-Seiwert S, Borkhardt A, Gierga K, Turowski B, Heiroth HJ, Steiger HJ, Stummer W. ALA-induced porphyrin accumulation in medulloblastoma and its use for fluorescence-guided surgery. Cent Eur Neurosurg. 2011 May;72(2):101-3. doi: 10.1055/s-0030-1252010. Epub 2010 Oct 7. No abstract available. PMID 20931449
- [Background] Foster N, Eljamel S. ALA-induced fluorescence image guided surgery of meningiomas: A meta-analyses. Photodiagnosis Photodyn Ther. 2016 Sep;15:73-8. doi: 10.1016/j.pdpdt.2016.05.006. Epub 2016 May 24. PMID 27235278
- [Background] Wainwright JV, Endo T, Cooper JB, Tominaga T, Schmidt MH. The role of 5-aminolevulinic acid in spinal tumor surgery: a review. J Neurooncol. 2019 Feb;141(3):575-584. doi: 10.1007/s11060-018-03080-0. Epub 2018 Dec 29. PMID 30594965
- [Background] Esteves S, Alves M, Castel-Branco M, Stummer W. A pilot cost-effectiveness analysis of treatments in newly diagnosed high-grade gliomas: the example of 5-aminolevulinic Acid compared with white-light surgery. Neurosurgery. 2015 May;76(5):552-62; discussion 562. doi: 10.1227/NEU.0000000000000673. PMID 25714513
- [Background] Lau D, Hervey-Jumper SL, Chang S, Molinaro AM, McDermott MW, Phillips JJ, Berger MS. A prospective Phase II clinical trial of 5-aminolevulinic acid to assess the correlation of intraoperative fluorescence intensity and degree of histologic cellularity during resection of high-grade gliomas. J Neurosurg. 2016 May;124(5):1300-9. doi: 10.3171/2015.5.JNS1577. Epub 2015 Nov 6. PMID 26544781
- [Background] Kaneko S, Kaneko S. Fluorescence-Guided Resection of Malignant Glioma with 5-ALA. Int J Biomed Imaging. 2016;2016:6135293. doi: 10.1155/2016/6135293. Epub 2016 Jun 27. PMID 27429612
- [Background] Cozzens JW, Lokaitis BC, Moore BE, Amin DV, Espinosa JA, MacGregor M, Michael AP, Jones BA. A Phase 1 Dose-Escalation Study of Oral 5-Aminolevulinic Acid in Adult Patients Undergoing Resection of a Newly Diagnosed or Recurrent High-Grade Glioma. Neurosurgery. 2017 Jul 1;81(1):46-55. doi: 10.1093/neuros/nyw182. PMID 28498936
- [Background] Acerbi F, Broggi M, Schebesch KM, Hohne J, Cavallo C, De Laurentis C, Eoli M, Anghileri E, Servida M, Boffano C, Pollo B, Schiariti M, Visintini S, Montomoli C, Bosio L, La Corte E, Broggi G, Brawanski A, Ferroli P. Fluorescein-Guided Surgery for Resection of High-Grade Gliomas: A Multicentric Prospective Phase II Study (FLUOGLIO). Clin Cancer Res. 2018 Jan 1;24(1):52-61. doi: 10.1158/1078-0432.CCR-17-1184. Epub 2017 Oct 10. PMID 29018053
- [Background] Kamp MA, Fischer I, Buhner J, Turowski B, Cornelius JF, Steiger HJ, Rapp M, Slotty PJ, Sabel M. 5-ALA fluorescence of cerebral metastases and its impact for the local-in-brain progression. Oncotarget. 2016 Oct 11;7(41):66776-66789. doi: 10.18632/oncotarget.11488. PMID 27564260
- [Background] Cornelius JF, Slotty PJ, El Khatib M, Giannakis A, Senger B, Steiger HJ. Enhancing the effect of 5-aminolevulinic acid based photodynamic therapy in human meningioma cells. Photodiagnosis Photodyn Ther. 2014 Mar;11(1):1-6. doi: 10.1016/j.pdpdt.2014.01.001. Epub 2014 Jan 31. PMID 24486853
- [Background] Della Puppa A, Rustemi O, Gioffre G, Troncon I, Lombardi G, Rolma G, Sergi M, Munari M, Cecchin D, Gardiman MP, Scienza R. Predictive value of intraoperative 5-aminolevulinic acid-induced fluorescence for detecting bone invasion in meningioma surgery. J Neurosurg. 2014 Apr;120(4):840-5. doi: 10.3171/2013.12.JNS131642. Epub 2014 Jan 10. PMID 24410157
- [Background] Widhalm G, Wolfsberger S, Minchev G, Woehrer A, Krssak M, Czech T, Prayer D, Asenbaum S, Hainfellner JA, Knosp E. 5-Aminolevulinic acid is a promising marker for detection of anaplastic foci in diffusely infiltrating gliomas with nonsignificant contrast enhancement. Cancer. 2010 Mar 15;116(6):1545-52. doi: 10.1002/cncr.24903. PMID 20108311
- [Background] Hendricks BK, Sanai N, Stummer W. Fluorescence-guided surgery with aminolevulinic acid for low-grade gliomas. J Neurooncol. 2019 Jan;141(1):13-18. doi: 10.1007/s11060-018-03026-6. Epub 2018 Oct 26. PMID 30367383
- [Background] Stummer W, Reulen HJ, Meinel T, Pichlmeier U, Schumacher W, Tonn JC, Rohde V, Oppel F, Turowski B, Woiciechowsky C, Franz K, Pietsch T; ALA-Glioma Study Group. Extent of resection and survival in glioblastoma multiforme: identification of and adjustment for bias. Neurosurgery. 2008 Mar;62(3):564-76; discussion 564-76. doi: 10.1227/01.neu.0000317304.31579.17. PMID 18425006
- [Background] Pichlmeier U, Bink A, Schackert G, Stummer W; ALA Glioma Study Group. Resection and survival in glioblastoma multiforme: an RTOG recursive partitioning analysis of ALA study patients. Neuro Oncol. 2008 Dec;10(6):1025-34. doi: 10.1215/15228517-2008-052. Epub 2008 Jul 30. PMID 18667747
- [Background] Stummer W, Tonn JC, Mehdorn HM, Nestler U, Franz K, Goetz C, Bink A, Pichlmeier U; ALA-Glioma Study Group. Counterbalancing risks and gains from extended resections in malignant glioma surgery: a supplemental analysis from the randomized 5-aminolevulinic acid glioma resection study. Clinical article. J Neurosurg. 2011 Mar;114(3):613-23. doi: 10.3171/2010.3.JNS097. Epub 2010 Apr 16. PMID 20397896
- [Background] Pineros M, Sierra MS, Izarzugaza MI, Forman D. Descriptive epidemiology of brain and central nervous system cancers in Central and South America. Cancer Epidemiol. 2016 Sep;44 Suppl 1:S141-S149. doi: 10.1016/j.canep.2016.04.007. PMID 27678316
- [Background] Sinning M, Frelinghuysen M, Gallegos M, Cordova A, Paredes P, Vogel C, Sujima E, Kamiya-Matsuoka C, Valdivia F. Outcome of patients with primary glioblastoma in Chile: single centre series. Ecancermedicalscience. 2021 Feb 10;15:1184. doi: 10.3332/ecancer.2021.1184. eCollection 2021. PMID 33777177